CLINICAL TRIAL: NCT05662111
Title: A Randomized, Placebo-controlled, Double-blind Trial to Study the Effects of Etidronate on Ectopic CALCIfication in FAhr's Disease or Syndrome
Brief Title: Treatment of Ectopic Calcification in Fahr's Disease or Syndrome
Acronym: CALCIFADE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands Brain Foundation (Other)
Responsible Party: Principal Investigator, H.L. Koek, MD, PhD, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL 83131.041.22; 2022-003299-17 (EudraCT Number); DR-2021-00387 (Other Grant/Funding Number: Hersenstichting)
Record Dates: First submitted 2022-11-16; First posted 2022-12-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Fahr Disease; Fahr Syndrome; Primary Familial Brain Calcification
MeSH Terms: conditions — Fahr's disease | interventions — Etidronic Acid

STUDY DESIGN:
Intervention Model Description: A randomized placebo-controlled double blind trial using etidronate versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Etidronate (Active Comparator): Etidronate 20 mg/kg for two weeks on and ten weeks off during 12 months
  Interventions: Drug: Etidronate
- Placebo (Placebo Comparator): Placebo for two weeks on and ten weeks off during 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etidronate — The dosage of etidronate is 20 mg/kg for twee weeks and ten weeks off. Etidronate is given in capsules of 200 mg. Etidronate capsules are administered orally. During the study, participants will receive etidronate in four periods of two weeks during the twelve months of follow-up.
  Other Names: Etidronate disodium
  Arms: Etidronate
Drug: Placebo — Placebo is given in capsules and are administered orally. During the study, participants will receive placebo in four periods of two weeks during the twelve months of follow-up.
  Other Names: Etidronate disodium
  Arms: Placebo

SUMMARY:
Fahr's disease or syndrome are neurodegenerative diseases in which patients present with bilateral vessel associated calcifications in the basal ganglia. The clinical penetration of Fahr's disease or syndrome is incomplete and heterogeneous comprising of neuropsychiatric signs, cognitive decline, movement disorders, and various other signs (migraine, speech disorders, pain, seizures). The symptoms start between 30 and 50 years and are (slowly) progressive. Symptomatic patients have an increased risk for dependence in activities of daily living and impaired quality of life.

Currently, disease-modifying therapies are not available for patients with Fahr's disease or syndrome. However, in a small case series it was shown that alendronate was effective in the clinical treatment of several patients with Fahr's disease or syndrome. Now the time has come to investigate the effectiveness of treatment with bisphosphonates in patients with Fahr's disease or syndrome in a randomized controlled trial.

DETAILED DESCRIPTION:
Fahr's disease, scientifically known as primary familial brain calcification (PFBC), is a neurodegenerative disease in which all patients present with bilateral vessel associated calcifications in the basal ganglia in the absence of other secondary causes of brain calcifications. When a secondary cause is identified, the term Fahr's syndrome is often used. Dominantly-inherited PFBC is associated with mutations in four genes; solute carrier family 20 member 2 (SLC20A2), xenotropic and polytropic retrovirus receptor 1 (XPR1), platelet-derived growth factor b (PDGFB) and platelet-derived growth factor receptor b (PDGFRB). Recessively inherited PFBC is associated with mutations in two genes; myogenesis-regulating glycosidase (MYORG) and junctional adhesion molecule 2 (JAM2). Mutations in the known genes account for half of patients, suggesting genetic heterogeneity, with new genes yet to be discovered. The estimated minimal prevalence in studies with PFBC diagnosed with genetic and imaging studies is 2.1 to 6.6 per 1,000 suggesting that PFBC is actually not a rare disorder and is underdiagnosed. The clinical penetration of Fahr's disease or syndrome is incomplete and heterogeneous comprising of neuropsychiatric signs (depression, anxiety, psychosis), cognitive decline, movement disorders (ataxia, dystonia, Parkinsonism) and various other signs (migraine, speech disorders, pain, seizures). The symptoms start between 30 and 50 years and are (slowly) progressive. Symptomatic patients have an increased risk for dependence in activities of daily living and impaired quality of life.

Histology shows small vessel and capillary calcifications, vascular insufficiency and blood-brain barrier damage. Neural pathology has been described and there are indications that calcifications could interfere with neural circuitry. It is not known how mutations in different genes lead to a common pathology. Yet PFBC belongs to a group of genetic diseases that due to different types of faulty phosphor metabolism leads to a shortage of inorganic pyrophosphate (PPi). PPi is the strongest inhibitor of ectopic calcification in the body. PPi can be replaced by etidronate, a stable molecular homologue of PPi and a well known bisphosphonate that has been used widely. Presently, the rare genetic diseases Pseudoxanthoma Elasticum (PXE), Generalized Arterial Calcification of Infancy (GACI) and Arterial Calcification due to Cluster of Designation 73 (CD73) deficiency (ACDC) are successfully treated with this medication. In PFBC, it was shown that due to mutations in the SLC20A2 gene the Pi Transporter 2 (PiT2) is compromised. The PiT2 transporter plays an important role in the maintenance of Pi homeostasis which is essential for adenosine triphosphate synthesis. Another mutation, XPR1 is responsible for phosphate efflux and mutations here lead to calcium deposition in endothelial cells. Recently, it was shown that mutations in the PDGFB and PDGFRB genes cause osteoblast like cells to mediate in the calcification process, as was also shown in PXE, GACI and ACDC patients.

Currently, disease-modifying therapies are not available for patients with Fahr's disease or syndrome. However, in a small case series it was shown that alendronate was effective in the clinical treatment of several patients with Fahr's disease or syndrome. Now the time has come to investigate the effectiveness of treatment with bisphosphonates in patients with Fahr's disease or syndrome in a randomized controlled trial.

ELIGIBILITY:
Inclusion criteria are:

1. Age of 18 years or over,
2. Clinical diagnosis of Fahr's disease or syndrome. No international accepted diagnostic criteria for Fahr's disease or syndrome exist yet. It is diagnosed mostly based on the clinical presentation. For the present study the following criteria are used:

   1. Clinical symptoms consistent with a clinical diagnosis of Fahr's disease or syndrome.
   2. Bilateral calcifications of the basal ganglia as seen on the computed tomography (CT) scan of the head. To rule out basal ganglia calcifications due to aging, a CT based calcification score will be used as proposed by Nicolas et al. Calcification is graded from 0 (no calcification) to 5 (serious and confluent) in specific locations of the brain; lenticular, caudate, thalamus nuclei, subcortical white matter, cortex, cerebellar hemispheres, vermis, midbrain, pons, and medulla. The total calcification score (ranging from 0 to 80) is obtained by adding all location-specific points, where a score higher than the age-specific threshold points at Fahr's disease or syndrome.

      Furthermore, the next criteria are supportive for the clinical diagnosis of PFBC:
   3. Frequently, the family history is consistent with autosomal dominant inheritance. A positive family history with at least one relative in the first or second degree with symptoms of PFBC is supportive for the clinical diagnosis of PFBC.
   4. The presence of a (likely) pathogenic mutation in one of the PFBC-related genes is supportive for the clinical diagnosis of PFBC. Mutations in up to now 4 known genes are associated with an autosomal dominant pattern of inheritance: solute carrier family 20 member 2 (SLC20A2) (OMIM#213600), xenotropic and polytropic retrovirus receptor 1 (XPR1) (OMIM#616413), platelet-derived growth factor b (PDGFB) (OMIM#615483), and platelet-derived growth factor receptor b (PDGFRB) (OMIM#615007). Autosomal recessively inherited PFBC is associated with mutations in two genes: myogenesis-regulating glycosidase (MYORG) (OMIM#618317) and junctional adhesion molecule 2 (JAM2) (OMIM#618824).

Exclusion criteria are:

1. unable or unwilling to sign an informed consent,
2. severe renal impairment (estimated glomerular filtration rate (eGFR) of <30 ml/min/1.73m2 calculated using CKD-EPI equation),
3. contraindication to receiving oral medication (for example severe dysphagia),
4. known abnormality of the oesophagus that would interfere with the passage of the drug (for example oesophageal strictures or achalasia),
5. known sensitivity to etidronate,
6. pregnancy, women with an active pregnancy wish <1 year, or women who are breastfeeding at the time of inclusion,
7. inability to undergo a Dutch neuropsychological assessment (for example, non-fluent Dutch speakers or severe visual, hearing or motor impairment),
8. any other medical or social condition that puts the subject at risk of harm during the study or might adversely affect the interpretation of the study data,
9. use of bisphosphonates during the last 5 years,
10. hypocalcaemia (calcium <2.20 mmol/L),
11. 25-OH vitamin D deficiency <35 nmol/L. After correction of hypocalcaemia or vitamin D deficiency, a participant is again suitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall cognitive functioning | 12 months
  Montreal Cognitive Assessment (MoCA; range 0-30, higher scores mean better outcome)
Memory | 12 months
  Composite z-score of Rivermead Behavioral Memory Test (RBMT) Stories immediate and delayed recall, Rey complex figure test immediate and delayed recall
Attention and speed of information processing | 12 months
  Composite z-score of Wechsler Adult Intelligence Scale third edition (WAIS-III) Digit Span Forward, Trail Making Test A (TMT-A), Stroop I and II
Executive functioning | 12 months
  Composite z-score of Wechsler Adult Intelligence Scale third edition (WAIS-III) Digit Span Backward, Trail Making Test B (TMT-B), Stroop III, semantic and letter fluency
Social cognition | 12 months
  Facial Expressions of Emotion - Stimuli and Tests (FEEST; scored based on normative data)

SECONDARY OUTCOMES:
Mobility | 12 months
  Condensed version of the Balance Evaluation Systems Test (Mini-BESTest), which is a composite test of gait and balance (range 0-28, higher scores mean better outcome)
Mobility | 12 months
  Unified Parkinson's Disease Rating Scale, part III (UPDRS; range 0-56, higher scores mean worse outcome)
Neuropsychiatric symptoms | 12 months
  Neuropsychiatric Inventory (NPI; range 0-144, higher scores mean worse outcome)
Activities of daily living | 12 months
  Katz-15 scale (range 0-15, higher scores mean worse outcome)
Quality of life questionnaire | 12 months
  36-item Short Form Health Survey (SF-36; range 0-100, higher scores mean better outcome)
Brain calcification volume | 12 months
  Volume of calcification quantified in computed tomography scan (milliliters)

CONTACTS AND LOCATIONS:
Overall Officials: Huiberdina L Koek, MD, PhD, Principal Investigator — UMC Utrecht
Locations (2):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers upon request. Due to the fact that Fahr's disease or syndrome is rare, not all data will be published openly, since this data might be traceable to an individual person.

REFERENCES:
- [Derived] Snijders BM, Mathijssen G, Peters MJ, Emmelot-Vonk MH, de Jong PA, Bakker S, Crommelin HA, Ruigrok YM, Brilstra EH, Schepers VP, Spiering W, van Valen E, Koek HL. The effects of etidronate on brain calcifications in Fahr's disease or syndrome: rationale and design of the randomised, placebo-controlled, double-blind CALCIFADE trial. Orphanet J Rare Dis. 2024 Feb 7;19(1):49. doi: 10.1186/s13023-024-03039-7. PMID 38326858